CLINICAL TRIAL: NCT07102979
Title: Remedial Mechanisms of Simvastatin and Ursodeoxycholic Acid in Liver Cirrhosis: Crosstalk Between Bile Secretion, Gut Microbiome, and Host Immune Response
Brief Title: Remedial Mechanism of Simvastatin and Ursodeoxycholic Acid in Liver Cirrhosis: Crosstalk of Bile Secretion, Gut Microbiome, and Host Immune Response
Acronym: SURGIC-Liver
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 202201398A3; CMRPG8P0291 (Other Grant/Funding Number: Chang Gung Memorial Hospital)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis; fecal bile salt; UDCA; statin
MeSH Terms: conditions — Liver Cirrhosis | interventions — Ursodeoxycholic Acid; Simvastatin

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, parallel-group study with four arms. Eligible participants with stable liver cirrhosis are randomly assigned in a 1:1:1:1 ratio to receive either (1) no treatment (control), (2) ursodeoxycholic acid (UDCA) alone, (3) simvastatin alone, or (4) a combination of simvastatin and UDCA for 6 months.
  Randomization is performed using block randomization to ensure balanced allocation across groups. The groups are followed in parallel, and no crossover occurs between arms. A separate healthy control group (non-cirrhotic) provides baseline microbiota and bile acid profile comparisons but is not included in the interventional randomization.
Masking Description: This is an open-label study. No participants, investigators, or outcome assessors are masked to treatment allocation. All parties involved are aware of the assigned interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Group (No Intervention): Participants receive standard clinical monitoring without any investigational treatment. No simvastatin or ursodeoxycholic acid (UDCA) is administered during the 6-month study period.
- UDCA Group (Experimental): Participants receive ursodeoxycholic acid (UDCA) at a dose of 10 mg/kg/day orally for 6 months to evaluate its effect on liver fibrosis, bile acid metabolism, and gut microbiota.
  Interventions: Drug: Simvastatin
- Simvastatin Group (Experimental): Participants receive simvastatin at a dose of 40 mg/day orally for 6 months. The treatment aims to assess effects on fibrosis markers, inflammation, and gut microbiota composition.
  Interventions: Drug: Ursodeoxycholic Acid (URSO)
- Simvastatin + UDCA Group (Experimental): Participants receive a combination of simvastatin (40 mg/day) and ursodeoxycholic acid (UDCA) (10 mg/kg/day) orally for 6 months. The combination therapy is evaluated for potential synergistic effects on fibrosis reduction, bile acid modulation, and microbiota restoration.
  Interventions: Drug: Ursodeoxycholic Acid (URSO); Drug: Simvastatin

INTERVENTIONS:
Drug: Ursodeoxycholic Acid (URSO) — Ursodeoxycholic acid (UDCA) was administered orally at a dose of 10 mg/kg/day for 6 months.
  Arms: Simvastatin + UDCA Group; Simvastatin Group
Drug: Simvastatin — Simvastatin was administered orally at a dose of 40 mg/day for 6 months.
  Arms: Simvastatin + UDCA Group; UDCA Group

SUMMARY:
The goal of this clinical trial is to learn whether simvastatin alone or in combination with ursodeoxycholic acid (UDCA) can reduce liver fibrosis, inflammation, and gut microbiota imbalance in patients with liver cirrhosis who have achieved viral eradication after hepatitis C or inactive hepatitis B.

The main questions the study aims to answer are:

Can simvastatin or UDCA reduce biomarkers of liver fibrosis and chronic inflammation?

Do these treatments improve gut microbiota composition and bile acid metabolism?

Is combination therapy more effective than either drug alone?

In this study, 120 patients with stable liver cirrhosis will be randomly assigned to one of four groups: no treatment (control), UDCA alone, simvastatin alone, or simvastatin plus UDCA. Patients will be followed for 6 months, during which stool, blood, and skin samples will be collected to assess gut microbiota, bile acid profiles, inflammatory markers, and fibrosis indicators.

A group of 30 healthy individuals without cirrhosis will also provide baseline comparisons for microbiota and bile acid profiles.

DETAILED DESCRIPTION:
Introduction There is emerging evidence that the gut milieu plays an important role in the progression of complications of cirrhosis. Studies have found dysbiosis in the gut microbiota in patients with cirrhosis, which has the potential to influence complications such as hepatic encephalopathy. The gut milieu in cirrhosis involves the interaction between the microbiota and secreted factors, such as bile acids (BAs), that can also modulate the gut barrier. The gut microbiota is known to convert primary bile acids - chenodeoxycholic acid (CDCA) and cholic acid (CA) - into the secondary bile acids lithocholic acid (LCA) and deoxycholic acid (DCA), respectively. Cirrhotic patients have been shown to have a lower proportion of secondary bile acids in their bile, although the mechanism for this remains unclear. Since bile acids have important downstream pathophysiologic effects, a better understanding of their interaction with the intestinal microbiome is crucial for gaining insight into the pathophysiology of cirrhosis.

In a previous study, the median abundances of certain microbial taxa were significantly altered in cirrhosis - with higher levels of Enterobacteriaceae and Veillonellaceae and lower levels of beneficial autochthonous bacteria such as Blautia, Ruminococcaceae, and Lachnospiraceae - especially in advanced cirrhosis compared to healthy controls. The total bile acid concentration in healthy stool was much higher than that in advanced cirrhosis, and secondary bile acids were significantly reduced in cirrhotic patients. Ratios of secondary to primary bile acids (e.g., DCA/CA and LCA/CDCA) were also lowest in advanced cirrhosis. The cirrhosis dysbiosis ratio (CDR) - defined as the ratio of beneficial to pathogenic bacteria - is significantly higher in healthy individuals and patients with compensated cirrhosis than in those with decompensated disease. A low CDR has been associated with increased risk of hepatic encephalopathy.

Bile acids are endogenous ligands for receptors such as Farnesoid X receptor (FXR), Takeda G protein receptor 5 (TGR5), and Sphingosine-1-phosphate receptor 2 (S1PR2). These receptors are located at the interface of the host immune system and gut microbiota and are abundantly expressed in cells of innate immunity, including intestinal and hepatic macrophages, dendritic cells, and natural killer T cells.

Ursodeoxycholic acid (UDCA) has been shown to enhance bile acid synthesis via CYP7A1 and to alter gut microbiota populations. It also has anticholestatic, antifibrotic, antiproliferative, and anti-inflammatory effects. Retrospective studies suggest that statins are safe in patients with compensated cirrhosis and may significantly reduce fibrosis. Preclinical models have demonstrated that statins improve endothelial function, reduce portal hypertension, and decrease fibrogenesis through pathways involving KLF2, eNOS, and other molecular targets. Animal studies further indicate that fluvastatin, lovastatin, and simvastatin inhibit hepatic stellate cell activation and reduce fibrotic signaling.

Statin therapy has also been associated with reduced prevalence of gut dysbiosis. The combination of UDCA and statins has been shown to be safe in humans and may have synergistic effects in lowering bile cholesterol levels. However, there is currently no prospective research evaluating whether this combination can improve fibrosis markers or gut microbial composition in cirrhotic patients.

Study Objective The primary objective of this study is to evaluate whether simvastatin alone or in combination with UDCA can reduce liver fibrosis markers, pro-inflammatory cytokines, and gut microbiota dysbiosis in patients with liver cirrhosis who have achieved viral eradication of chronic hepatitis C or have undetectable viral load in hepatitis B.

Study Design and Population We aim to enroll 120 stable patients at a single center who have achieved a sustained virologic response (SVR) after hepatitis C treatment or maintained undetectable hepatitis B viral load for at least 6 months. Eligible patients must have been diagnosed with liver cirrhosis (FIB-4 ≥ 3.25) and meet Baveno VII criteria (liver stiffness measurement [LSM] ≥ 25 kPa). Patients with LSM < 15 kPa and platelet count ≥ 150 × 10⁹/L will be excluded. The Baveno VII "grey zone" will be stratified into high-risk and low-risk categories based on LSM and platelet counts.

Exclusion criteria include: current statin use, diabetes mellitus, liver cancer, alcoholic liver disease, moderate-to-severe fatty liver, decompensated cirrhosis (jaundice, ascites, hepatic encephalopathy, esophageal/gastric varices), chronic kidney disease, recent antibiotic use (within 3 months), and ongoing use of proton pump inhibitors.

Participants will be randomly assigned into four groups (n = 30 per group):

Group 1: Control (no intervention)

Group 2: UDCA (10 mg/kg/day)

Group 3: Simvastatin (40 mg/day)

Group 4: Simvastatin (40 mg/day) + UDCA (10 mg/kg/day)

Samples will be collected at baseline and after 6 months of treatment, including fecal samples (for microbiota and bile acid profiles), skin bile acid swabs, inflammatory cytokine levels, and serum fibrosis biomarkers. Non-invasive liver stiffness measurements will also be performed.

In addition, 30 non-cirrhotic patients (FIB-4 < 1.45) who have achieved SVR after hepatitis C treatment will serve as a healthy comparator group for microbiota and bile acid analysis.

Randomization Block randomization will be used. Eligible patients will be assigned in a 1:1:1:1 ratio using a block of 8 with two patients per group.

Microbiota and Bile Acid Analysis Stool samples will be processed using standardized DNA extraction methods. 16S rRNA gene sequencing (targeting the V4 region) will be performed, followed by bioinformatic analysis. Bile acids in fecal and skin samples will be analyzed using LC-MS/MS and TD-ESI/MS techniques, respectively.

Primary Outcome Change in fibrosis biomarkers (TGF-β1, Type IV collagen, hyaluronic acid, and FIB-4 Index) from baseline to 6 months.

Secondary Outcomes Change in cirrhosis dysbiosis ratio (CDR)

Change in total and secondary/primary fecal bile acid ratios

Change in serum inflammatory cytokines (IL-6, IL-8, IL-10, TNF-α)

Sample Size Justification There are currently no prospective data available to determine the optimal sample size for evaluating changes in fibrosis with simvastatin and UDCA. Previous studies evaluating simvastatin's effect on portal pressure included 24 patients per arm and reported a significant HVPG reduction. Based on this, 30 participants per group have been selected to ensure adequate power.

Safety Monitoring Simvastatin will start at 20 mg/day and may be increased to 40 mg/day after 4 weeks if tolerated. Creatine kinase and liver function tests will be checked after 2 weeks. Adverse events and side effects will be recorded throughout the study. Statins have been shown to be safe in patients with chronic liver disease, with low reported risk of adverse events and a potential reduction in all-cause mortality.

Statistical Analysis Risks will be reported as incidence rate ratios (IRRs) with 95% confidence intervals and p-values. Subgroup analyses and interaction tests will be performed. Time-to-event data will be analyzed using life-table methods and log-rank tests. A p-value < 0.05 will be considered statistically significant. Analyses will be performed using SAS version 9.1.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years
* Diagnosed with primary liver cirrhosis (FIB-4 ≥ 3.25)
* Liver stiffness measurement (LSM) ≥ 25 kPa, or classified into the Baveno VII "grey zone"
* Achieved sustained virological response (SVR) at least 6 months after hepatitis C treatment, or
* Non-replicating hepatitis B infection (undetectable viral load) for at least 6 months
* Able and willing to provide informed consent

Exclusion Criteria:

* Current or prior use of statins
* Liver decompensation (jaundice, ascites, hepatic coma, or esophagogastric varices)
* Diagnosed hepatocellular carcinoma or other liver cancers
* Alcoholic liver disease or moderate-to-severe fatty liver
* Diagnosed diabetes mellitus
* Chronic kidney disease
* Use of antibiotics within the past 3 months
* Use of gastric ulcer medications such as proton pump inhibitors (PPIs)
* Pregnancy or breastfeeding
* Any condition deemed by the investigator to interfere with study participation or outcomes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in liver fibrosis biomarker (TGF-β1) | Baseline and 6 months after treatment initiation
  Measurement of serum fibrosis-related marker TGF-β1. This will assess the antifibrotic effects of simvastatin, UDCA, and their combination in patients with stable liver cirrhosis.
Change in liver fibrosis biomarker (Type IV collage) | Baseline and 6 months after treatment initiation
  Measurement of serum fibrosis-related marker Type IV collagen. This will assess the antifibrotic effects of simvastatin, UDCA, and their combination in patients with stable liver cirrhosis.
Change in liver fibrosis biomarker (Hyaluronic Acid) | Baseline and 6 months after treatment initiation
  Measurement of serum fibrosis-related marker Hyaluronic Acid. This will assess the antifibrotic effects of simvastatin, UDCA, and their combination in patients with stable liver cirrhosis.
Change in liver fibrosis biomarker (FIB-4 Index) | Baseline and 6 months after treatment initiation
  Measurement of serum fibrosis-related marker FIB-4 Index.. This will assess the antifibrotic effects of simvastatin, UDCA, and their combination in patients with stable liver cirrhosis.

SECONDARY OUTCOMES:
Change in Cirrhosis Dysbiosis Ratio (CDR) | Baseline and 6 months after treatment
  CDR is calculated as the ratio of beneficial autochthonous bacteria (e.g., Lachnospiraceae, Ruminococcaceae, Clostridiales) to potentially pathogenic bacteria (e.g., Enterobacteriaceae, Streptococcaceae), using 16S rRNA sequencing of stool samples.
Change in Serum Inflammatory Cytokines | Baseline and 6 months after treatment
  Measurement of circulating cytokines including IL-6, IL-8, IL-10, and TNF-α to evaluate systemic inflammatory response to intervention.
Change in Skin Bile Acid Profile | Baseline and 6 months after treatment
  Quantitative analysis of bile acid composition on skin surface using TD-ESI/MS to explore systemic bile acid signaling and excretion pathways.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Others, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to privacy concerns and data protection regulations. The study does not have participant consent or institutional approval for public data sharing. Aggregated results will be reported in scientific publications.

REFERENCES:
- [Result] Islam KB, Fukiya S, Hagio M, Fujii N, Ishizuka S, Ooka T, Ogura Y, Hayashi T, Yokota A. Bile acid is a host factor that regulates the composition of the cecal microbiota in rats. Gastroenterology. 2011 Nov;141(5):1773-81. doi: 10.1053/j.gastro.2011.07.046. Epub 2011 Aug 10. PMID 21839040
- [Result] Chen Y, Yang F, Lu H, Wang B, Chen Y, Lei D, Wang Y, Zhu B, Li L. Characterization of fecal microbial communities in patients with liver cirrhosis. Hepatology. 2011 Aug;54(2):562-72. doi: 10.1002/hep.24423. Epub 2011 Jun 26. PMID 21574172
- [Result] Bajaj JS, Hylemon PB, Ridlon JM, Heuman DM, Daita K, White MB, Monteith P, Noble NA, Sikaroodi M, Gillevet PM. Colonic mucosal microbiome differs from stool microbiome in cirrhosis and hepatic encephalopathy and is linked to cognition and inflammation. Am J Physiol Gastrointest Liver Physiol. 2012 Sep 15;303(6):G675-85. doi: 10.1152/ajpgi.00152.2012. Epub 2012 Jul 19. PMID 22821944
- [Result] Bajaj JS, Ridlon JM, Hylemon PB, Thacker LR, Heuman DM, Smith S, Sikaroodi M, Gillevet PM. Linkage of gut microbiome with cognition in hepatic encephalopathy. Am J Physiol Gastrointest Liver Physiol. 2012 Jan 1;302(1):G168-75. doi: 10.1152/ajpgi.00190.2011. Epub 2011 Sep 22. PMID 21940902

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT07102979/Prot_ICF_000.pdf